CLINICAL TRIAL: NCT02653378
Title: The Effects of Acute Caloric Deprivation on Odour Identification and Food Reward
Acronym: DEXDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Eric Doucet, Professor of Human Kinetics, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H09-09-03
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Olfaction; Diet; Exercise; Energy Depletion; Food Hedonics; Food Reward
MeSH Terms: conditions — Anosmia; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DIET ARM (Active Comparator): A 25% energy depletion (daily for 3 days) induced by reducing the amount of energy intake that would otherwise keep the individual in energy balance.
  Interventions: Behavioral: DIET
- EX ARM (Active Comparator): A 25% energy depletion (daily for 3 days) induced by performing aerobic exercise at 50% of V02max.
  Interventions: Behavioral: EX

INTERVENTIONS:
Behavioral: DIET — 25% Energy Depletion by Diet only for 3 Days
  Arms: DIET ARM
Behavioral: EX — 25% Energy Depletion by Exercise only for 3 Days
  Arms: EX ARM

SUMMARY:
The purpose of this study is to determine how the modality of energy depletion can differently impact appetite hormones, ad libitum food intake, food hedonics, and olfaction.

DETAILED DESCRIPTION:
The objectives of the current randomized controlled study were to examine how the modality of an acute 3 day isocaloric -25% energy depletion by dieting alone or by aerobic exercise alone differently impacts appetite and appetite-related hormones, ad libitum energy intake (EI), food hedonics and food reward, and olfaction. It was hypothesized that independent of modality of depletion, that relative to the control, there would be increased ad libitum feeding and food reward, improvements in smell performance, and a decline in fasting leptin and increase in fasting total ghrelin. It was also hypothesized that the increased food reward would prove to be a predictor of ad libitum EI and that relative to the depletion by aerobic exercise alone, the depletion by diet alone would produce greater compensatory increases in appetite, ad libitum EI, and food reward.

Statistics

To test for differences in body weight, plasma hormone concentrations, relative-reinforcing value of food (RRVF), and olfaction across each condition of the study, repeated measures ANOVA controlling for day 1 as a covariate was employed. Pairwise comparisons at day 4 using Sidak adjustment to account for multiple comparisons are reported when the ANOVA was significant. One way repeated measures ANOVAs with Sidak adjustments for multiple comparisons were used to test for differences in variables measured only at day 4: body composition (fat mas, %Fat, and fat free mass), appetite, palatability, and ad libitum EI.

ELIGIBILITY:
Inclusion Criteria:

* Free from any illness that could influence outcome of the experiment
* Weight-stable for >6months
* aged between 18-40 years

Exclusion Criteria:

* diabetic
* smoker
* medication

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in Ad Libitum Energy Intake at Buffet Lunch--total kcals consumed at lunch meal measured to nearest 0.5grams. | Day 1 and Day 4 of each study arm (DIET and EX)
  Ad libitum measure of energy intake at lunch time at Day 1 and Day 4 of study

SECONDARY OUTCOMES:
Change in fasting measure of Leptin | Day 1 and Day 4 of each study arm (DIET and EX)
  One fasting sample of plasma Leptin
Change in fasting measure of Ghrelin | Day 1 and Day 4 of each study arm (DIET and EX)
  One fasting sample of plasma Ghrelin taken at Day 1 and Day 4 of study
Change in Relative-Reinforcing Value of Food as measured by food points earned during a computerized behavioral choice tast | Day 1 and Day 4 of each study arm (DIET and EX)
  Computer task measuring reinforcing value of preferred snack food and preferred fruit at Day 1 and Day 4 of study
Olfaction--Odor Detection Threshold measured by Sniffin Sticks odorized pens | Day 1 and Day 4 of each study arm (DIET and EX)
  Measure of odour threshold for n-butanol taken at Day 1 and Day 4 of study

CONTACTS AND LOCATIONS:
Overall Officials: Eric Doucet, PhD, Principal Investigator — University of Ottawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McNeil J, Lamothe G, Cameron JD, Riou ME, Cadieux S, Lafreniere J, Goldfield G, Willbond S, Prud'homme D, Doucet E. Investigating predictors of eating: is resting metabolic rate really the strongest proxy of energy intake? Am J Clin Nutr. 2017 Nov;106(5):1206-1212. doi: 10.3945/ajcn.117.153718. Epub 2017 Sep 6. PMID 28877891
- [Derived] Cameron JD, Goldfield GS, Riou ME, Finlayson GS, Blundell JE, Doucet E. Energy depletion by diet or aerobic exercise alone: impact of energy deficit modality on appetite parameters. Am J Clin Nutr. 2016 Apr;103(4):1008-16. doi: 10.3945/ajcn.115.115584. Epub 2016 Feb 17. PMID 26888712